CLINICAL TRIAL: NCT03599752
Title: The Role of Multimodality Management in Risk-Stratified Patients With Lung-Limited Metastatic Colorectal Cancer
Brief Title: Chemotherapy and/or Metastasectomy in Treating Patients With Metastatic Colorectal Adenocarcinoma With Lung Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0905; NCI-2018-01456 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0905 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Adenocarcinoma; Colorectal Carcinoma Metastatic in the Lung; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Metastasectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1A (chemotherapy, metastasectomy) (Experimental): Low risk patients receive standard of care chemotherapy for 3 months prior to and 3 months after undergoing metastasectomy in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Chemotherapy; Procedure: Metastasectomy
- Group 1B (metastasectomy) (Experimental): Low risk patients undergo metastasectomy.
  Interventions: Procedure: Metastasectomy
- Group 2A (metastasectomy) (Experimental): High risk patients undergo metastasectomy.
  Interventions: Procedure: Metastasectomy
- Group 2B (chemotherapy) (Experimental): High risk patients continue standard of care chemotherapy for 6 months in the absence of disease progression or unacceptable toxicity. Patients with stable disease or radiographic response after 6 months may then cross over to Group 2A.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Receive chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
  Arms: Group 1A (chemotherapy, metastasectomy); Group 2B (chemotherapy)
Procedure: Metastasectomy — Undergo pulmonary metastasectomy
  Arms: Group 1A (chemotherapy, metastasectomy); Group 1B (metastasectomy); Group 2A (metastasectomy)

SUMMARY:
This phase II trial studies how well chemotherapy and/or metastasectomy work in treating patients with colorectal adenocarcinoma that has spread to the lungs (metastases). Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Metastasectomy is a surgical procedure that removes tumors formed from cells that have spread from other places in the body. It is not yet known if chemotherapy and metastasectomy together works better in treating patients with metastatic colorectal adenocarcinoma with lung metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare recurrence-free survival in patients with "low risk" lung-limited metastatic colorectal cancer (mCRC) undergoing pulmonary metastasectomy with or without perioperative chemotherapy.

II. To compare overall survival in patients with "high risk" lung-limited mCRC receiving systemic chemotherapy with or without surgical resection.

SECONDARY OBJECTIVES:

I. To compare grade 3 and 4 adverse events in patients receiving surgical resection and/or chemotherapy in the management of lung-limited mCRC.

EXPLORATORY OBJECTIVES:

I. To evaluate for changes in circulating tumor deoxyribonucleic acid (DNA) following surgical resection and/or systemic chemotherapy in patients with lung-limited mCRC.

OUTLINE: Patients are assigned to 1 of 2 risk groups (low or high).

GROUP 1 (LOW RISK): Patients are randomized to 1 of 2 groups.

GROUP 1A: Patients receive standard of care chemotherapy for 3 months prior to and 3 months after undergoing metastasectomy in the absence of disease progression or unacceptable toxicity.

GROUP 1B: Patients undergo metastasectomy.

GROUP 2 (HIGH RISK): All high risk patients receive standard of care chemotherapy for 3 months in the absence of disease progression or unacceptable toxicity. Patients without progressive disease after 3 months are then randomized to 1 of 2 groups.

GROUP 2A: Patients undergo metastasectomy.

GROUP 2B: Patients continue standard of care chemotherapy for 6 months in the absence of disease progression or unacceptable toxicity. Patients with stable disease or radiographic response after 6 months may then cross over to Group 2A.

After completion of study treatment, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of colorectal adenocarcinoma
* Metastatic colorectal cancer involving the lung classified as determined by the treating clinical team
* Diagnosis of colorectal metastasis to lung made either histologically with trans-thoracic needle biopsy or clinically based on radiographic imaging
* Identification as a medically appropriate candidate for surgical resection of the lung metastasis (metastases) according to the evaluating cardiothoracic surgeon. Standard justification for deeming a patient medically operable based on:

  * Pulmonary reserve adequate to tolerate complete resection of all intrathoracic disease, as deemed by thoracic surgeon, which may be determined by:

    * Baseline forced expiratory volume in one second (FEV1) > 40% predicted
    * Post-operative predicted FEV1 > 30% predicted
    * Diffusion capacity of the lung for carbon monoxide (DLCO) > 40% predicted
    * Absent baseline hypoxemia and/or hypercapnia
    * Exercise oxygen consumption > 50% predicted
    * Absent severe pulmonary hypertension
    * Absent severe cerebral, cardiac, or peripheral vascular disease
    * Absent severe chronic heart disease
  * Ability to tolerate surgical resection and acceptable operative risk as deemed by thoracic surgeon based on performance status and medical comorbidities
* Identification as a medically appropriate candidate for systemic chemotherapy at the discretion of the evaluating medical oncologist
* Resection/definitive therapy of primary colorectal tumor with no suspicion of recurrence. Prior radiation to a rectal adenocarcinoma is permitted
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Ability to provide informed consent for participation
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Hemoglobin >= 9.0 gm/dL
* Platelet count >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (except patients with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Serum creatinine =< 1.5 x ULN OR creatinine clearance (CrCl >= 50 mL/min (if using the Cockcroft-Gault formula)
* Patients (men and women) of child bearing potential should use an effective (for them) method of birth control throughout their participation in this study

Exclusion Criteria:

* Tumor involvement at other metastatic sites (e.g., liver, distant lymph nodes) that has not been definitively treated. Prior surgical resection for metastatic disease at other (non-pulmonary) sites is permitted
* Presence of intact primary colorectal adenocarcinoma (or of an anastomotic recurrence)
* Previous radiotherapy to a lung metastasis that is still detectable radiographically
* Known dihydropyrimidine dehydrogenase (DPD) deficiency that would preclude the patient from tolerating 5- fluorouracil chemotherapy
* Prior intolerance of systemic therapies used as standard regimens in the treatment of metastatic CRC that would prohibit further receipt of systemic chemotherapy and/or biologic agents -e.g.,5-fluorouracil, oxaliplatin, irinotecan, anti-VEGF therapies (e.g., bevacizumab, ramucirumab), or anti-EGFR therapies (e.g., cetuximab, panitumumab, for patients with RAS wild-type colorectal tumors)
* Prior therapy with regorafenib or trifluridine/tipiracil (TAS-102) for metastatic/unresectable colorectal cancer
* Synchronous primary or prior malignancy in the past 5 years other than non-melanomatous skin cancer or in situ cancer
* Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (Low risk) | Up to 2 years
  The primary objective for the low risk group is to evaluate the efficacy of chemotherapy plus surgical resection versus surgical resection alone measured by recurrence-free survival (RFS). The event includes recurrence and death due to any cause. Patients will be stratified at randomization according to three variables: age (age >= 60 years vs age < 60 years), RAS mutation status (mutant vs wild type), and location of primary tumor within colon/rectum (right/cecum/ascending colon/hepatic flexure/transverse colon vs left/distal to transverse colon).
Overall survival (High risk) | Up to 2 years
  The primary objective for the high-risk group is to evaluate the efficacy of chemotherapy plus surgical resection versus chemotherapy alone measured by overall survival (OS). The event includes death due to any cause. Patients will be stratified at randomization according to 4 variables: response to chemotherapy in the preceding three months of treatment (complete or partial response vs stable disease by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria), RAS mutated vs RAS wild type tumors, right versus left-sided primary tumors, and oxaliplatin-based vs irinotecan-based chemotherapy in the initial treatment period on study.

CONTACTS AND LOCATIONS:
Overall Officials: Mara B. Antonoff, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (4):
  - Washington University School of Medicine, St Louis, Missouri
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Baylor Colllege of Medicine, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
- Canada (2):
  - University Health Network Princess Margaret Cancer Center P2C, Toronto, Ontario
  - University of Montreal, Montreal, Quebec

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org